CLINICAL TRIAL: NCT03365245
Title: Partial Least Squares Regression Modelling for Glaucoma Detection Using Retinal Nerve Fiber Layer, Ganglion Cell Layer and Visual Field Data
Brief Title: Partial Least Squares Regression Modelling for Glaucoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PLSR
Record Dates: First submitted 2017-11-04; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Visual Field Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Other): Microperimetry and automated visual field are performed at three different days
  Interventions: Device: Microperimetry; Device: automated visual field

INTERVENTIONS:
Device: Microperimetry — Microperimetry is performed at three different days
Device: automated visual field — Automated visual field ist performed at three different days

SUMMARY:
A partial least squares regression model for visual field testing among glaucoma patients will be developed.

In addition, microperimetry will be compared to conventional perimetry and reproducibility will be assessed.

DETAILED DESCRIPTION:
Aim of this study is to develop a partial least squares regression model incorporating retinal nerve fiber layer (RNFL) and retinal ganglion cell layer (RGCL) measurements as well as visual field testing to represent a glaucoma expert opinion on the stage of glaucoma.

In addition, microperimetry will be compared to conventional perimetry and reproducibility will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* written informed consent prior to surgery
* any glaucoma-associated changes in one or both eyes (i.e. increased intraocular pressure, optic disc changes, known visual field defects) in the "glaucoma patients" and the absence of any glaucoma associated changes in the "healthy eyes group".

Exclusion Criteria:

* Secondary glaucoma
* In case of pregnancy (pregnancy test will be taken in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
partial least square regression | one month
  Development of a partial least squares regression model to detect glaucoma

SECONDARY OUTCOMES:
reproducibility | one month
  Comparison of reproducibility of microperimetry and visual field testing
Retinal nerve fiber thickness (RNFL) and the the retinal ganglion cell layer (RGCL) | one month
  The retinal nerve fiber layer thickness and the thickness of the retinal ganglion cell layer will be compared
Microperimetry versus visual field testing | one month
  Comparison of microperimetry and visual field testing

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS, Vienna, Austria